CLINICAL TRIAL: NCT00423865
Title: A Phase I Study of Weekly Low-Dose Cisplatin Plus Escalating Doses of Oral RAD001(Everolimus) for Patients With Advanced Solid Tumors
Brief Title: Cisplatin and Everolimus in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSKCC 06-129; MSKCC-06129; NCT00406666 (obsolete NCT alias)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2012-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; CISPLATIN; RAD001 (EVEROLIMUS); 06-129
MeSH Terms: interventions — Cisplatin; Everolimus; Gene Expression Profiling; Immunohistochemistry; Biopsy

ARMS (1):
- cisplatin & RAD001 (Experimental): This will be a single institution phase I study of low dose weekly cisplatin (20 mg/m2 intravenously on Days 1, 8, and 15) plus escalating doses of daily RAD001 tablets (per oral or via percutaneous gastrostomy tube, Days 1 -21 of a 28-Day Cycle) for patients with advanced solid tumors
  Interventions: Drug: cisplatin; Drug: everolimus; Genetic: gene expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: biopsy

INTERVENTIONS:
Drug: cisplatin — cisplatin (20 mg/m2 intravenously on Days 1, 8, and 15)
Drug: everolimus — escalating doses of daily RAD001 tablets (per oral or via percutaneous gastrostomy tube, Days 1 -21 of a 28-Day Cycle)
Genetic: gene expression analysis — Each biopsy specimen will be formalin-fixed and paraffin-embedded for IHC, and analysis of p53 and p21 will follow methods previous reported by our group. The avidin-biotin immunoperoxidase technique will be employed.
Other: immunohistochemistry staining method — After the phase 2 recommended dose is established in the phase I portion of the study (Part A), we plan to enroll an additional 6 patients for pharmacodynamic studies (Part B). Entry into Part B requires the patient have tumor tissue which is easily accessible for research biopsy. The patients will be asked to provide written informed consent for the research biopsies. Patients also will be asked to provide written informed consent to allow the use of their tissue for future research studies. The research biopsies are not mandatory for any patient. Patients who do not consent to the research biopsies or who withdraw consent for the research biopsies may still receive RAD001 + cisplatin in the study
Other: laboratory biomarker analysis — Laboratory data (complete blood count, comprehensive metabolic panel including magnesium) regarding adverse events will be collected on each cisplatin treatment day. Additional adverse event data will be collected at regularly scheduled clinic visits at which history and physical are performed by the investigator (Cycle 1 - Days 1, 8, 15, and 21. Cycle 2 - Days 1 and 15. Cycle 3 and beyond - Day 1)
Other: pharmacological study — For patients in Part A, research bloods for pharmacokinetics are drawn on Day 1 and Day 8.
Procedure: biopsy — "Pre-treatment Research Biopsy:" Within 14 days prior to treatment, research biopsy (of primary tumor, metastatic deposit, or involved lymph node) will be performed. Baseline labs should be drawn within 14 days of the research biopsy. The biopsy sample will be formalin-fixed and paraffin-embedded for immunohistochemistry. Post-treatment Research Biopsy:" Research biopsy (of primary tumor, metastatic deposit, or involved lymph node) will be requested again for Day 15 of Cycle 1, prior to administration of RAD001 and cisplatin on that day.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Everolimus may also help cisplatin work better by making tumor cells more sensitive to the drug. Giving cisplatin together with everolimus may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with cisplatin in treating patients with advanced solid tumors or recurrent or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended phase II dose of everolimus when administered with low-dose cisplatin in patients with advanced solid tumors.

Secondary

* Determine the safety and tolerability of this regimen in these patients.
* Describe the pharmacokinetics of this regimen in patients with advanced solid tumors.
* Assess the effects of this regimen on p53 and p21 immunohistochemistry assays of pre- and post-treatment tumor biopsies from patients with recurrent or metastatic solid tumors.

OUTLINE: This is a dose-escalation study of everolimus (part A) followed by a biological marker study (part B).

* Part A (closed to accrual as of 1/2009): Patients receive cisplatin* IV over 30 minutes on days 1, 8, and 15 and oral everolimus* once daily on days 1-21. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose proceeding that at which 2 of 6 patients experience dose-limiting toxicity (DLT) during course 1. The recommended phase II dose is defined as the dose at which 1 of 6 patients experience DLT during course 1.

Blood is drawn periodically on days 1 and 8 of course 1 for pharmacokinetic studies.

* NOTE: *Patients who have completed 5 courses of treatment and maintain stable disease or better may continue treatment with everolimus alone or in combination with cisplatin
* Part B: Patients undergo biopsy of the primary tumor, metastatic deposit, or involved lymph node. No more than 14 days later, patients receive everolimus at the recommended phase II dose and cisplatin as in part A.

Patients undergo another tumor biopsy on day 15 of course 1, before receiving chemotherapy. The pre- and post-therapy tissue is examined by immunochemistry and analyzed for p53 and p21 expression.

PROJECTED ACCRUAL: A total of 30 people will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Advanced solid tumor (part A)

    * Confirmation by core biopsy or fine-needle aspiration allowed
  * Solid tumor (part B)

    * Recurrent or metastatic disease
    * Easily accessible for biopsy
* Measurable disease
* No uncontrolled brain or leptomeningeal metastases

  * No requirement for glucocorticoids

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin > 10 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (< 5 times ULN if liver metastases are present)
* Creatinine normal OR creatinine clearance ≥ 55 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after completion of study therapy
* No HIV positivity
* No peripheral neuropathy ≥ grade 2
* No hypertriglyceridemia ≥ grade 2
* No impaired gastrointestinal function or gastrointestinal disease that may alter the absorption of everolimus, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea
  * Vomiting
  * Diarrhea
  * Malabsorption syndrome
  * Small bowel resection
* No other concurrent severe and/or uncontrolled medical disease that would compromise study participation, including any of the following:

  * Uncontrolled diabetes
  * Unstable angina
  * New York Heart Association class III or IV congestive heart failure

PRIOR CONCURRENT THERAPY:

* No more than 3 prior cytotoxic chemotherapy regimens for recurrent or metastatic disease
* At least 4 weeks since prior major surgery and recovered
* At least 4 weeks since prior radiation therapy and recovered
* At least 4 weeks since prior systemic anticancer therapy and recovered
* At least 4 weeks since prior and no other concurrent investigational drugs
* No prior everolimus or other agents specifically targeting mTOR
* No prior radiation therapy to > 25% of the bone marrow
* No prior radiation therapy to the whole pelvis and/or brain
* No concurrent chronic steroid treatment (> 5 mg/day of prednisone)

  * Concurrent low-dose steroid replacement regimens (≤ 5 mg/day of prednisone) allowed
* No concurrent immunosuppressive agents
* No other concurrent anticancer agents
* No concurrent agents known to be strong inhibitors or inducers of isoenzyme CYP3A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of everolimus | 1 year

SECONDARY OUTCOMES:
Pharmacokinetic profile of cisplatin and everolimus | 1 year
Pharmacodynamic profile of cisplatin and everolimus | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew G. Fury, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; David G. Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States